CLINICAL TRIAL: NCT06380660
Title: A Phase I/II, Open-label, Multicentre Study to Assess the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Preliminary Efficacy of Ascending Doses of ACE-86225106 as Monotherapy in Patients With Advanced Solid Tumors
Brief Title: Study of ACE-86225106 to Treat Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Acerand Therapeutics (Shanghai) Limited (Industry)
Responsible Party: Sponsor
Organization: Acerand Therapeutics Limited (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACE-106-001
Record Dates: First submitted 2024-04-16; First posted 2024-04-24 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Solid Tumor, Adult; BRCA1 Mutation; BRCA2 Mutation; Ovarian Cancer; Breast Cancer; Prostate Cancer
Keywords: ACE-86225106; advanced solid tumors; PARP inhibitor; BRCA mutation; breast cancer; ovarian cancer; CRPC
MeSH Terms: conditions — Ovarian Neoplasms; Breast Neoplasms; Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ACE-86225106 tablet (Experimental): ACE-86225106 tablet monotherapy
  Interventions: Drug: ACE-86225106 tablet

INTERVENTIONS:
Drug: ACE-86225106 tablet — ACE-86225106 will be administered orally daily as a continuous regimen. Subjects will continue to receive study treatment until PD as judged by local investigator review, development of unacceptable toxicity, or withdrawal of consent.

SUMMARY:
The purpose of this study is to determine if the experimental treatment with poly-ADP ribose polymerase (PARP) inhibitor, ACE-86225106 is safe, tolerable and has anti-cancer activity in adult patients with advanced solid tumors.

DETAILED DESCRIPTION:
This study is a Phase I/II, open-label, multicentre study of ACE-86225106 administered orally in patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent;
2. Advanced solid tumors, difficult to treat or intolerant to standard treatment, suitable for investigational treatment;
3. Has Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1;
4. Has a life expectancy of at least 3 months;
5. Has measurable disease per RECIST 1.1, castration-resistant prostate Ccancer (CRPC) patients can be assessed according to PCWG3;
6. Adequate organ function and bone marrow function;
7. Can provide tumor specimens and blood samples for Homologous Recombination Deficiency (HRD)/ Homologous Recombination Repair (HRR) related gene testing.

Exclusion Criteria:

1. Receiving any anti-cancer drugs, major surgery, extensive radiation therapy, or local radiation therapy within protocol-defined wash-out period;
2. Concomitant use of medications or herbal supplements known to be strong or moderate inhibitors or inducers of cytochrome P450 3A4 (CYP3A4);
3. Receiving continuous corticosteroid treatment with a dose of prednisone greater than 10 mg/day or an equivalent dose.
4. Receiving continuous treatment with prednisone at a dose of >10 mg/d or other corticosteroids at an equivalent dose for any reason.
5. Any previous treatment-related toxicities have not recovered, i.e., to ≤ Grade 1 (as evaluated by NCI-CTCAE v5), except alopecia and other Grade 2 toxicities that are deemed not to affect the conduct of the study, as assessed by the sponsor and the clinical investigator.
6. Spinal cord compression or brain metastases unless asymptomatic, treated and stable.
7. Severe cardiovascular disorders.
8. Myelodysplastic syndrome (MDS)/acute myeloid leukemia (AML) or with evidence suggesting possible MDS/AML.
9. Concomitant diseases or conditions that would preclude the absorption of the investigational product.
10. Active infections, or a known history of HIV infection, or a known active hepatitis B or C, or a known active tuberculosis.
11. Other malignancies that require treatment within 3 years prior to first dose of study investigational product.
12. Conditions with rapid deterioration during the screening period.
13. Known allergy or hypersensitivity to the investigational product or any of the excipients of the investigational product.
14. Has other medical conditions that at the discretion of investigator interfere with safety or efficacy evaluation, or affect treatment compliance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 298 (Estimated)
Dates: Start 2024-03-22 (Actual); Primary Completion 2028-12-21 (Estimated); Study Completion 2029-03-21 (Estimated)

PRIMARY OUTCOMES:
Number of participants experiencing adverse events (AEs)/serious adverse events (SAEs) | From time of information consent to 30 days post last dose, up to 3 years
  Number of participants with incidence of adverse events and with serious adverse events including changes from baseline in laboratory parameters, vital signs, ECGs, and physical examination, etc.
The number of patients experiencing dose limiting toxicity (DLT), as defined in the protocol | From the first dose of ACE-86225106 on Cycle 1 Day 1 up to and including the planned end of Cycle 1 (at the end of 28 days)
  A DLT is defined as any toxicity events related to ACE-86225106 that occur from the first dose of study treatment until the planned end date of Cycle 1 (DLT assessment period), meeting the criteria specified in protocol.
Recommended Phase 2 dose (RP2D) and/or maximum tolerated dose (MTD) | Up to 3 years
  RP2D will be finally determined by the Safety Monitoring Committee (SMC) and sponsor based on all data from the dose escalation module and backfill module, as well as the exposure-response relationship evaluated (if available). MTD is defined as the maximum dose level at which ≤1 patient have DLTs during the DLT observation period, and it should be determined with 6 evaluable patients.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to 3 years
  ORR is defined as proportion of patients who achieved complete response (CR) or partial response (PR) according to RECIST 1.1 recorded from first investigational product treatment until disease progression or death due to any cause. The confirmation of response for patients who has PR or CR at first time should be performed by at least 4 weeks. For castration-resistant prostate cancer (CRPC) patients, bone lesion will be assessed according to PCWG3 criteria.
Duration of Response (DoR) and Time to Response (TTR) | Up to 3 years
  DOR is defined, for patients with an objective response, as the time from first documentation of objective tumor response (CR or PR) to the first documentation of objective tumor progression or death due to any cause.
Progression Free Survival (PFS) | Up to 3 years
  PFS is defined as the time from the first study treatment to the date of the first documentation of objective progression of disease (PD) or death due to any cause.
Overall Survival (OS) | Up to 3 years
  OS is defined as the time from the first study treatment to the date of death due to any cause
Pharmacokinetic (PK) parameters and Pharmacodynamic (PD) marker change | Up to 3 years
  Blood drug concentrations at each scheduled time point will be summarized descriptively, and individual and mean concentration-time curves will be plotted by dose group.
Serum tumor marker change: CA125, etc. (OC), prostatic specific antigen (PSA, prostate cancer) decreased, and specific tumor markers for other tumor types may also be included (to be assessed by clinical investigators) | Up to 3 years
  The tests for the above serum tumor markers will support the tumor response evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Sherwin Cai, MD, Study Director — Acerand Therapeutics
Locations (14):
- China (14):
  - Chongqing Cancer Hospital, Chongqing, Chongqing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong
  - Anyang Cancer Hospital, Anyang, Henan
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - Jinan Central Hospital, Jinan, Shandong
  - Qilu Hospital Shangdong University, Jinan, Shandong
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Second Hospital Affiliated to Shanxi Medical University, Taiyuan, Shanxi
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - First Hospital Affiliated to Wenzhou Medical University, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No